CLINICAL TRIAL: NCT00585403
Title: PBMC, Exercise and Children: Initial Mechanisms
Brief Title: Exercise Changes to Peripheral Blood Mononuclear Cells in Children
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: PBMC Exercise [2004-3967]; HL-80947
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Physical Fitness; Obesity; Child Development; Growth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells, plasma, serum, mRNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children: Early and late pubertal girls and boys

SUMMARY:
The goal of this research is to determine how the peripheral immune system is altered by exercise and differences related to gender, pubertal status and health.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

1. To systematically measure for the first time in healthy children and adolescents the effects of brief bouts of exercise on:

   1. Numbers of circulating PMBCs, their subsets and key intercellular adhesion molecules (ICAMs).
   2. PBMC gene regulation of stress, inflammatory, and growth/repair mediators [including: interleukin-4 (IL-4), IL-6, IL-10, tumor necrosis factor-alpha (TNF-alpha), interferon-gamma), growth hormone (GH), insulin-like growth factor-I (IGF-I), heat shock proteins (Hsp)].
   3. Circulating (serum) and intracellular PBMC levels of key mediators by flow cytometry and cell culture techniques.
   4. Circulating endogenous triggers of PBMC mediator responses-soluble Hsp, IL-6, and F2-isoprostanes.
2. To determine how the acute PBMC responses are altered by gender, pubertal status, body composition (measured by whole-body and regional DEXA), and fitness (measured by progressive cycle ergometry and gas exchange).
3. To determine the relationship in healthy children and adolescents among acute PBMC responses to exercise, biochemical precursors of the metabolic syndrome (insulin, glucose, lipids), and the balance of the TH1/TH2 immune response.

ELIGIBILITY:
Inclusion Criteria:

* appropriate Tanner Stage
* No evidence of disease or disability

Exclusion Criteria:

* no use of antiinflammatory medications, alcohol, illegal drugs or bronchodilators
* elite children participating in extensive exercise or dance programs
* pregnant

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Early and late pubertal boys and girls recruited from Orange County, CA
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan M Cooper, M.D., Principal Investigator — Univ. California, Irvine, CA
Locations (1):
- General Clinical Research Center, Orange, California, United States